CLINICAL TRIAL: NCT01022476
Title: A Pilot Study of Pharmacokinetics, Tolerance and Efficacy of Raltegravir Combined to Two Fully Active Molecules Among Nucleosi(ti)de Analogs and Enfuvirtide Before and After Liver Transplant in HIV Infected Patients With End Stage Liver Disease (ANRS 148 LIVERAL)
Brief Title: Raltegravir in Patients With End Stage Liver Disease and in Transplant Recipients
Acronym: LIVERAL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-014616-36; ANRS 148 LIVERAL (Other: ANRS)
Record Dates: First submitted 2009-11-26; First posted 2009-12-01 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2013-07

CONDITIONS: HIV Infection; Liver Failure; Evidence of Liver Transplantation
Keywords: Pharmacokinetics; Raltegravir; Immunosuppressive Agents; Severe hepatic insufficiency; Liver Transplantation; Additional Keywords; HIV Infection; Hepatocarcinoma; Hepatitis C; Hepatitis B
MeSH Terms: conditions — HIV Infections; Liver Failure; Hepatic Insufficiency; Carcinoma, Hepatocellular; Hepatitis C; Hepatitis B | interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Raltegravir potassium (Experimental): raltegravir 400 mg twice a day
  Interventions: Drug: Raltegravir potassium

INTERVENTIONS:
Drug: Raltegravir potassium — one pill of raltegravir 400 mg twice a day
  Other Names: ISENTRESS

SUMMARY:
This phase I/II, multi-center study is designed to determine the pharmacokinetic profile of Raltegravir in patients with end stage liver disease and to assess drug-drug interaction when Raltegravir is combined with immunosuppressive therapy in liver transplant recipients.

DETAILED DESCRIPTION:
HIV infected patients with stable plasma HIV-RNA below 50 copies per mL and severe liver dysfunction will be switched from their antiretroviral regimen to a combination of raltegravir (one 400 mg pill twice daily) and two fully active molecules among nucleosi(ti)de analogs and enfuvirtide for a first period of at least 3 months and a second period of at least 3 months after liver transplantation, if need be, when a steady state of the anticalcineurin will be reached. Pharmacokinetic parameters of raltegravir will be calculated during severe liver dysfunction period and after liver transplantation. Pharmacokinetic parameters of cyclosporine (or tacrolimus if contra indication to cyclosporine) will be compared when administrated alone or combined with raltegravir. Patients will be followed up according to standard of care. This study will be divided in two distinct periods (1 and 2) lasting 3 months each. Period 1 will start from the inclusion in the study and will generally include the switch to raltegravir. Period 2 will start from liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Documented HIV-1 infection, hepatitis B or C co-infection is allowed
* Plasma viral load at screening visit below 50 copies per mL for at least 6 months
* Patient with severe liver failure (Meld Score ≥ 15 and/or refractory ascites and/or haemorrhage of digestive tract and/or hepatic encephalopathy) for taking part into period 1
* Patient eligible for the liver transplant waiting list or immediate post transplantation for taking part into period 2
* Abstinence from alcohol intake for at least 6 months (WHO norm)
* Withdrawal from intravenous drug use for at least 6 months (methadone substitution is permitted)
* No ongoing class C opportunistic infection (1993 CDC classification)
* Patient whose clinical and immunovirological condition allows triple therapy with raltegravir + 2 NRTI or raltegravir + NRTI + enfuvirtide
* Patient whose HIV population, according to cumulative genotypes carried out on viral RNA together with treatment history (if available and interpreted as per the ANRS-AC11 algorithm version no.19) does not present a profile of mutations associated with resistance to raltegravir and is sensitive to at least two fully active* agents selected among nucleoside/nucleotide reverse transcriptase analogs NRTI (abacavir, lamivudine, emtricitabine, tenofovir) or enfuvirtide

  *An ARV agent is considered to be fully active if the cumulative genotypes do not show any mutation associated with resistance or any mutation associated with "possible resistance"
* Patient not having experienced viral escape during treatment combining 3TC, FTC or raltegravir
* Patient registered with or covered by a social security scheme
* For women of child-bearing potential, use of a barrier contraceptive method during sexual intercourse and negative pregnancy test (plasma ß-HCG ) at screening visit
* Informed consent form signed at screening visit at the latest

Exclusion Criteria:

* More than two virological failures during antiretroviral treatment
* Currently receiving treatment with an agent in development (apart from an authorization for temporary use)
* Plasma viral load at screening visit ≥ 50 copies per mL during at least the last 6 months
* Pregnant women, or women liable to become pregnant, breast-feeding women, no contraception, or refusal to use contraception
* All conditions (including but not limited to alcohol intake and drug use) liable to compromise, in the investigator's opinion, the safety of treatment and/or the patient's compliance with the protocol
* Patient not having any effective options for NRTI +/- enfuvirtide (defined in the inclusion criteria)
* Ongoing treatment with interferon-alpha or ribavirin for hepatitis C
* Concomitant medication including one or more agents liable to induce UGT1A1 and reduce raltegravir concentrations:

  * anti-infective agents: rifampicin/rifampin
  * psychotropic/antiepileptic agents: phenytoin, phenobarbital, carbamazepine
  * steroidal anti-inflammatory drug: dexamethasone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters of raltegravir in patients with severe liver dysfunction and after a liver transplantation when combined to immunosuppressive therapy. Pharmacokinetic parameters of immunosuppressive drugs with or without raltegravir | at month 1 for period 1 and day 7-month 1 for period 2

SECONDARY OUTCOMES:
To assess the maintenance of the virological efficacy on HIV of raltegravir combined with two fully active molecules among NRTI (or NRTI + enfuvirtide). Follow-up over a 3-months period before and after transplantation | from day 0 to month 3 for period 1 and period 2
To assess the safety of raltegravir before transplantation in patients with impaired liver function, and after transplantation in combination with immunosuppressive treatment | from day 0 to month 3 for period 1 and period 2
To describe the clinical outcome of patients (such as the onset of opportunistic infections, relapse of HCV infection, morphological and metabolic disorders outcomes) | from day 0 to month 3 for period 1 and period 2
To describe the changes in liver function (evaluation of liver function during treatment) before and after liver transplantation | from day 0 to month 3 for period 1 and period 2

CONTACTS AND LOCATIONS:
Overall Officials: Elina TEICHER, MD, Principal Investigator — Hôpital de Bicêtre - LE KREMLIN-BICETRE - FRANCE; Jean-Pierre ABOULKER, MD, Study Chair — INSERM SC10 VILLEJUIF FRANCE
Locations (1):
- Service de Médecine Interne, Hôpital de Bicêtre, Le Kremlin-Bicêtre, France

REFERENCES:
- See also: Agence nationale de recherches sur le sida et les hépatites virales — http://www.anrs.fr/